CLINICAL TRIAL: NCT00378235
Title: Phase I/II Trial of Intracerebral IL13-PE38QQR Infusions in Pediatric Patients With Recurrent Malignant Glioma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: There was a change of sponsor. The new sponsor company did not wish to conduct the study after all.
Sponsor: INSYS Therapeutics Inc (Industry)
Collaborators: Pediatric Brain Tumor Consortium (PBTC), St. Jude Children's Research Hospital (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL13PEI-151; NCI Protocol No.: PBTC-011
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Recurrent Malignant Glioma
Keywords: neurosurgery, craniotomy; convection-enhanced delivery; CNS interstitial infusion; recombinant toxins; malignant glioma, recurrent; catheter,; intratumoral therapy; positive pressure microinfusion
MeSH Terms: conditions — Glioma; Recurrence | interventions — IL13-PE38

INTERVENTIONS:
Drug: IL13-PE38QQR

SUMMARY:
IL13-PE38QQR is an oncology drug product consisting of IL13 (interleukin-13) and PE38QQR (a bacteria toxin). IL3-PE38QQR is a protein that exhibits cell killing activity against a variety of IL13-receptor positive tumor cell lines indicating that it may show a therapeutic benefit. In reciprocal competition experiments, the interaction between IL13-PE38QQR and the IL13 receptors was shown to be highly specific for human glioma cells.

DETAILED DESCRIPTION:
PHASE I OBJECTIVES:

I. To describe toxicities and estimate the maximum safe flow rate and maximum tolerated infusion concentration, of IL13-PE38QQR delivered after surgical resection by peritumoral infusion via 2 to 4 catheters positioned in the brain adjacent to the resection cavity, from the start of infusion through the DLT observation period.

II. To determine the IL13 receptor alpha-2 chain expression status and distribution in pediatric recurrent or progressive malignant gliomas.

III. To describe the overall safety and tolerability of IL13PE38QQR infusion from the start of infusion through disease progression or initiation of alternative treatment.

PHASE II OBJECTIVES:

I. To estimate the survival distribution post initial progression, at the maximum safe total flow rate and MTiC established in phase I.

II. To estimate the progression-free survival distribution for patients post-initial progression or recurrence at the maximum safe total flow rate and MTiC established in phase I.

III. To determine the serum levels of IL13-PE38QQR and distribution in pediatric recurrent or progressive malignant gliomas.

IV. To describe the overall safety and tolerability of IL13-PE38QQR infusion from the start of infusion through disease progression or initiation of alternative treatment.

PROTOCOL OUTLINE: At study entry, all patients will be registered prior to planned gross total resection (> 95% resection of the solid, contrast enhancing tumor component). On the day of catheter placement (CP, 2-7 days after resection), if the patient is neurologically stable, 2-4 catheters will be stereotactically placed. On day 1 after catheter placement, infusion of IL3-PE38QQR will begin if the patient is neurologically stable and will continue for 96 hours. In Phase I, the total flow rate and the concentration of IL3-PE38QQR will be determined by the dose escalation plan. In the Phase II evaluations of safety and efficacy, patients will be treated at the flow rate and concentration identified in Phase I.

PROJECTED ACCRUAL: Approximately 24 patients will participate in the Phase I portion of the study. During the Phase I portion, the rate-limiting factor is the time the study must be closed during the toxicity assessment period. Although it is estimated that 1.5 patients per month will enroll in the Phase I portion, the observed rate may be lower due to temporary suspensions in accrual. It is not possible to estimate the time required to complete the Phase I portion of the trial. It is estimated that approximately 26 patients will contribute to the Phase II portion. Using the same rough estimate of accrual, the Phase II portion may last about 3 years.

ELIGIBILITY:
-Disease Characteristics-

Must be at least 3 years but not more than 21 years of age.

Must have had surgery (or biopsy) of a supratentorial brain tumor with pathologic diagnosis of malignant (grade 3 or 4) glioma, including anaplastic astrocytoma, mixed anaplastic astrocytoma, or glioblastoma multiforme.

Must have radiographic evidence of recurrent or progressive supratentorial malignant glioma compared with a prior imaging study. The baseline tumor measurements must be determined within 2 weeks prior to study entry.

The tumor must have a solid component at least 1.0 cm in diameter.

Gross total resection must be planned, with the intent of removing all contrast-enhancing components of the tumor.

Must have received external beam radiotherapy, with tumor dose of at least 48 Gy; and must be completed at least 8 weeks prior to study entry.

-Patient Characteristics-

Karnofsky Performance Score for patients older than 16 years, or the Lansky Performance Scale for patients 16 years old or younger, must be at least 60.

Hematologic status: Absolute neutrophils at least 1,500/mm3; Hemoglobin at least 10 gm/dL (transfusion independent); Platelets at least 100,000/mm3 (transfusion independent); PT & aPTT less than or equal to the institutional upper limit of normal.

Must have recovered from toxicity of prior therapy: at least 6 months after Gliadel® wafer; at least 8 weeks after hematopoietic stem cell transplant; at least 4 weeks after any cytotoxic chemotherapy or any systemic investigational agent; at least 6 weeks after nitrosoureas; at least 2 weeks after vincristine or non-cytotoxic chemotherapy.

Patient's legal guardian must understand the investigational nature of this study and its potential risks and benefits; must sign informed consent.

No pregnant or breast-feeding patients. All patients of child-bearing age, male and female, must practice an effective method of birth control during the study.

No patients with multi-focal tumor not amenable to gross total resection or tumor dissemination (subependymal or leptomeningeal).

No patients with clinically significant increased intracranial pressure (e.g., impending herniation) uncontrolled seizures, or requirement for immediate palliative treatment.

No patients who received any localized antitumor therapy for the malignant glioma, either intracerebral chemotherapy (other than Gliadel®) or focal radiation therapy (e.g., stereotactic radiosurgery or brachytherapy).

No patients who are receiving concurrent chemotherapy (other than steroids) or any other investigational agent.

No patients unwilling to follow protocol requirements.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Banerjee, MD, MPH, Principal Investigator — University of California at San Francisco
Locations (10):
- United States (10):
  - University of California San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital, Chicago, Illinois
  - Dana-Farber Cancer Institute-Dept of Pediatric Oncology, Boston, Massachusetts
  - Duke University Medical Center-Dept. of Pediatrics, Medicine & Surgery, Durham, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine-Dept of Pediatrics, Houston, Texas
  - Children's Hospital & Regional Medical Center, Seattle, Washington